CLINICAL TRIAL: NCT03243188
Title: Palliative Care in General Practice: Cancer Patients' and Carers' Experience of Their General Practitioner's (GP's) Role
Brief Title: Palliative Care in General Practice: Cancer Patient/Carer Experience
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS ID 225027
Record Dates: First submitted 2017-07-27; First posted 2017-08-08 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2017-07

CONDITIONS: Cancer
Keywords: Palliative Care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Cancer patients with palliative care needs (+/- their carers)
  Interventions: Other: Qualitative interview

INTERVENTIONS:
Other: Qualitative interview — Qualitative data will be obtained through semi-structured interviews with adults with cancer and palliative care needs. Patients will be invited to bring their carer to the interview. EG will conduct and transcribe up to 30 audio-recorded semi-structured interviews, which will be carried out at the patient's preferred location (either at home, over the phone, or in a pre-booked room at St Joseph's Hospice). EG will ask questions relating to sociodemographic data (recording this on the Personal Information Sheet) prior to starting the interview.

SUMMARY:
Study Title: Palliative care in general practice: cancer patients' and carers' experience of their GP's role

Study Design: Qualitative interview study

Study Participants: Adult patients with cancer and palliative care needs, accompanied by their carers

Planned Sample Size: Up to 30 interviews with patients +/- their carers

Planned Study Period: October 2017 - December 2018

Research Question: What experience do adults with cancer, and carers, have of their GP's involvement in palliative care provision?

DETAILED DESCRIPTION:
Participants will be invited and recruited to the study from St Joseph's Hospice in Hackney (single centre study). Patients with cancer that are either attending the day centre service at St Joseph's or being visited at home by the community specialist palliative care nursing/medical team based at St Joseph's Hospice; will be approached by their direct clinical care staff. (Some of the direct clinical care team are National Health Service (NHS) staff and some care is commissioned by the NHS despite St Joseph's Hospice being a non-NHS site). Staff will initiate discussion about the project, and will assess for both mental and physical capacity to participate.

Dr Emilie Green (EG) will then contact the potential participants by phone or in person (if they have previously given verbal consent for her to join their usual clinical staff on a home visit or when they are attending the day centre). The project will be discussed with each potential participant, and EG will answer any questions they may have, will assess for mental and physical capacity, and will arrange a mutually convenient time and location to meet for the interview.

Before starting the interview, EG will again make time to clarify any questions each participant may have. She will ask each participant to date/sign three consent forms before starting the interview (one for EG, one for the participant, and one for their notes at St Joseph's Hospice). If a joint interview is undertaken with a patient and their carer; both parties will individually sign their own consent forms. She will then ask questions relating to sociodemographic data (recording this on the Personal Information Sheet) e.g. age, living situation and diagnosis before starting the interview. The interviews will each last at least 30 minutes.

If participants decide that they would like a telephone interview, the process will be slightly different. EG will send three consent forms to each prospective participant (one for them to keep, and two for them to date/sign and send back by post) in a stamped addressed envelope. If the forms are not received within 3 weeks, EG will follow up with a phone call to the prospective participant, to clarify whether they still wish to participate. Only after she receives the two dated/signed consent forms will EG arrange a time with them for the telephone interview. She will then phone the participant from a private location that she does not share with other colleagues. She will collect sociodemographic information (which will be recorded on the Personal Information Sheet) before starting the interview (which will last at least 30 minutes.)

Qualitative data will be obtained through semi-structured interviews with adults with cancer and palliative care needs. Patients will be invited to bring their carer to the interview. EG will conduct and transcribe up to 30 audio-recorded semi-structured interviews, which will be carried out at the patient's preferred location (either at home, over the phone, or in a pre-booked room at St Joseph's Hospice). EG will ask questions relating to sociodemographic data (recording this on the Personal Information Sheet) prior to starting the interview.

EG will transcribe all interviews verbatim. Data will be analysed thematically and will adhere to the principles of the Framework Analysis developed by Ritchie and Spencer. Recurring themes and concepts will be identified using a constant comparative approach. Any contributions made by carers will be included and analysed as 'added value' data.This will enable us to explore if and how carers' perspectives contribute to our understanding of patient experience of their GP's involvement in palliative care.

ELIGIBILITY:
Inclusion criteria for participants

* Patients either attending the St Joseph's Hospice day centre or being visited at home by their community specialist palliative care nursing/medical team and their carers
* Adult patients with a cancer diagnosis and their carers
* Able to understand and communicate in written and spoken English
* With mental and physical capacity to consent Exclusion criteria for participants
* Paediatric patients
* Patients without a cancer diagnosis
* Unable to understand written or spoken English
* Without mental and physical capacity to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be invited and recruited to the study from St Joseph's Hospice in Hackney (single centre study). Patients and their carers from all three geographical areas, served by St Joseph's, will be invited to participate: City & Hackney, Tower Hamlets and Newham. The Principal Investigator Jane Naismith (JN) working at St Joseph's Hospice will assist with and coordinate the recruitment process.
  This setting was chosen as it permits access to a varied group of patients and carers. A purposive sampling will ensure recruitment of patients across a breadth of socio-demographics, cancer diagnoses and experience of different GP practices.
  A target sample size of up to 30 interviews has been chosen, taking into account available time and resources.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
To explore the experience/perspectives of adults with cancer, and carers, of the role of their GP in providing palliative care, using a qualitative semi-structured interview schedule | October 2017 - December 2018
  To explore patients' and carers' experience of:
  1. The role of the GP in providing palliative care to adult patients with cancer
  2. The facilitators and barriers to the GP's capacity to fulfill this perceived role

CONTACTS AND LOCATIONS:
Overall Officials: Jane Naismith, Principal Investigator — St Joseph's Hospice; Patrick White, Study Director — King's College London; Heidi Lempp, Study Director — King's College London
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No